CLINICAL TRIAL: NCT05683171
Title: A Phase 1/2, Open-label Study of Valemetostat in Combination With Rituximab and Lenalidomide in Relapsed or Refractory Follicular Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0551; NCI-2023-00072 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 Dose Escalation (Experimental): The dose escalation phase will assess the safety/tolerability of escalating doses of valemetostat and lenalidomide when combined with rituximab
  Interventions: Drug: Rituximab; Drug: Lenalidomide; Drug: Valemetostat

INTERVENTIONS:
Drug: Rituximab — Given by IV (vein)
  Other Names: Rituxan
Drug: Lenalidomide — Given by PO
  Other Names: CC-5013; Revlimid™
Drug: Valemetostat — Given by PO

SUMMARY:
To find a recommended dose of valemetostat that can be given in combination with rituximab and lenalidomide to patients with follicular lymphoma. The safety and effects of this drug combination will also be studied

DETAILED DESCRIPTION:
Primary Objectives: Phase 1

--Evaluate the safety and tolerability of valemetostat in combination with R2 in subjects with R/R FL and determine the recommended phase 2 dose (RP2D) for evaluation in phase 2.

Secondary Objectives: Phase 1

* Evaluate the efficacy of valemetostat in combination with R2 in R/R FL
* Evaluate the pharmacokinetics (PK) of valemetostat in combination with R2

Exploratory Objective: Phase 1

* Evaluate pharmacodynamic profile of valemetostat
* Evaluate the efficacy of valemetostat in combination with R2 in R/R FL

Primary Objective: Phase 2

--Evaluate the efficacy of valemetostat in combination with R2 in R/R FL

Secondary Objective: Phase 2

* Evaluate the ORR
* Evaluate the DOR
* Evaluate the time to next anti-lymphoma treatment (TTNT)
* Evaluate the safety and tolerability
* Evaluate the PK of valemetostat in combination with R2

Exploratory Objective: Phase 2

* Evaluate the PFS of valemetostat in combination with R2 in R/R FL
* Evaluate OS
* Evaluate the effect of valemetostat in combination with R2 in R/R FL on epigenetic remodeling and gene expression
* Evaluate changes in tumor/immune microenvironment
* Evaluate pharmacodynamic profile of valemetostat

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the eligibility criteria to be enrolled on this study.

1. Subjects ≥18 years of age at the time the ICF is signed.
2. Have histologically confirmed FL, grades 1-3A
3. Must have been previously treated with at least 1 prior systemic therapy followed by relapsed, refractory or progressive disease.

   a. Systemic therapy includes: i. Anti-CD20 monoclonal antibody in combination with chemotherapy ii. Anti-CD20 monoclonal antibody monotherapy iii. Anti-CD20 monoclonal antibody in combination with lenalidomide iv. Anti-CD20 monoclonal antibody plus investigational agent on protocol
4. Requiring systemic therapy as assessed by investigator based on tumor size, location, and/or GELF criteria.
5. Bi-dimensionally measurable disease, with at least one mass lesion ≥ 2 cm in longest diameter by CT, PET/CT, and/or MRI which was not previously irradiated.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
7. Adequate renal function defined as calculated creatinine clearance per the Cockcroft and Gault formula

   * In phase 1, creatinine clearance must be >60 mL/minute
   * In Phase 2, creatinine clearance must be ≥30 mL/minute.
8. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC) ≥1,000/mm3 (≥1.0 × 109/L) if no lymphoma infiltration of bone marrow OR ANC ≥750/mm3 (≥0.75 × 109/L) with bone marrow infiltration, without growth factor support (filgrastim or pegfilgrastim) for at least 14 days.
   2. Platelet ≥75,000/mm3 (≥75 × 109/L). Evaluated at least 7 days after platelet transfusion.
   3. Hemoglobin > 8.0 g/dL. Evaluated at least 7 days after RBC transfusion.
9. Adequate liver function:

   1. Total bilirubin ≤1.5 × the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome (eg, a gene mutation in UGT1A1), who can have total bilirubin <3.0 mg/dL.
   2. ALT and AST ≤3 × ULN.
10. International normalized ratio (INR) ≤1.5 × ULN and activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless on warfarin, then INR ≤3.0).
11. If the subject is a female of childbearing potential, she must have a negative serum pregnancy test at Screening and must be willing to use 1 highly effective method and 1 additional effective birth control method upon enrollment, during the Treatment Period, and for 3 months, following the last dose of study drug. A female is considered of childbearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy) with surgery at least 1 month before the first dose of study drug or confirmed by follicle stimulating hormone (FSH) test >40 mIU/mL and estradiol < 40 pg/mL (<140 pmol/L).
12. If the subject is a male, the subject must be surgically sterile or willing to use a highly effective birth control upon enrollment, during the treatment period, and for 3 months following the last dose of study drug. Male subjects must not freeze or donate sperm starting at Screening and throughout the study period, and for at least 3 months after the final study drug administration
13. Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 3 months after the final study drug administration. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
14. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
15. Able and willing to provide written informed consent and to comply with the study protocol

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry.

1. Transformation to DLBCL at study entry
2. Grade 3B FL
3. Prior systemic therapy (eg, chemotherapy, immunomodulatory therapy, or monoclonal antibody therapy) within 3 weeks prior to the first dose of study drug.
4. Having progressive disease while on prior lenalidomide, discontinuing lenalidomide due to unacceptable toxicity, or prior lenalidomide therapy within the past 12 months prior to the first dose of study drug
5. Had curative radiation therapy or major surgery within 4 weeks or palliative radiation therapy within 2 weeks prior to the first dose of study drug
6. Systemic treatment with corticosteroids (>10 mg daily prednisone equivalents). Note: Short-course systemic corticosteroids (eg, prevention/treatment for transfusion reaction) or use for a non-cancer indication (eg, adrenal replacement) is permissible
7. History of autologous stem cell transplant within 60 days prior to first dose of study drug
8. History of allogeneic stem cell transplant within 90 days prior to the first dose of study drug, and clinically significant graft-versus-host disease (GVHD) or GVHD requiring systemic immunosuppressive prophylaxis or treatment
9. Prior malignancy active within the previous 2 years except for locally curable cancer that is currently considered as cured, such as cutaneous basal or squamous cell carcinoma, superficial bladder cancer, or cervical carcinoma in situ, or an incidental histological finding of prostate cancer
10. Presence or history of central nervous system (CNS) involvement of lymphoma
11. Prior EZH inhibitor therapy
12. Current use of moderate or strong cytochrome P450 (CYP)3A inducers (See Appendix E) or inhibitors, or prior use of moderate or strong CYP3A within the past 2 weeks.
13. Current use of P-gp inducers and on narrow therapeutic index, sensitive P-gp substrates.
14. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of lenalidomide capsules, or put the study outcomes at undue risk
15. Human immunodeficiency virus (HIV), active Hepatitis C Virus, active Hepatitis B Virus infection, or any active systemic infection. Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated.
16. Clinically significant cardiovascular disease such asymptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
17. Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block. QT prolongation is not a significant ECG abnormality that would warrant exclusion.
18. Lactating or pregnant subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Nastoupil, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org